CLINICAL TRIAL: NCT06903598
Title: Anesthesia and Analgesia Methods in Pediatric External Ventricular Drainage Placement
Brief Title: Scalp Blocks for Pediatric External Ventricular Drainage Placement
Status: Completed | Type: Observational
Sponsor: Hande Gurbuz (Other Government)
Collaborators: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Sponsor-Investigator, Hande Gurbuz, Assoc. Prof., MD, PhD, Bursa City Hospital
Organization: Bursa City Hospital (Other Government)
Other Study IDs: 2011-KAEK-25 2021/08-24
Record Dates: First submitted 2025-03-24; First posted 2025-03-31 (Actual); Last update posted 2025-03-31 (Actual); Status verified 2025-03

CONDITIONS: Hydrocephalus in Children; Regional Block; Pediatric Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Scalp Block: Those who underwent surgery with scalp block
- Local infiltration: Those who underwent surgery with local anesthetic infiltration

SUMMARY:
External ventricular drainage (EVD) provides cerebrospinal fluid drainage in hydrocephalus. In adults, the neurosurgeon can place EVD at the bedside. In children, it is mainly preferred to be placed in the operating room under general anesthesia. However, general anesthesia may negatively affect oxygenation (during the intubation period) or cerebral blood flow (due to hypotension). This study investigates the use of regional block methods (without general anesthesia) in children for EVD placement.

DETAILED DESCRIPTION:
External ventricular drainage (EVD) provides cerebrospinal fluid drainage in hydrocephalus. In adults, EVD can be placed by the neurosurgeon at the bedside. In children, it is mainly preferred to be placed in the operating room under general anesthesia. However, general anesthesia may negatively affect oxygenation during a prolonged intubation period, leading to hypoxemia. Furthermore, hypotensive effects of general anesthesia may cause ischemia due to decreased cerebral blood flow.

Additionally, on the other hand, painful stimuli caused by surgical incisions or pins may cause hemorrhagic events due to a hypertensive period. Therefore, scalp blocks and local anesthetic infiltrations are recommended to prevent such adverse events. Although general anesthesia has been a routine for many anesthesiologists for EVD placement in children, this research hypothesizes that scalp blocks (along with sedatives) can be used as an anesthesia method for EVD placement.

This study investigates the use of regional block methods (to avoid general anesthesia) in children for EVD placement.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing external ventricular drainage

Exclusion Criteria:

* Children who were intubated preoperatively.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under 18 undergoing external ventricular drainage placement in the operating room between 2021 and 2022 in Bursa Yuksek Ihtisas TRH.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2021-08-25 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Anesthesia method | From enrollment to the end of surgery
  The anesthesia method used for the surgery (general anesthesia or sedation)

SECONDARY OUTCOMES:
Analgesic consumption | Postoperative first 24 hours.
  Total analgesic consumption within the first 24 in the postoperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Yildirim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The data sets used in this research may be made available upon reasonable request to the corresponding author.

REFERENCES:
- [Background] Rigamonti A, Garavaglia MM, Ma K, Crescini C, Mistry N, Thorpe K, Cusimano MD, Das S, Hare GMT, Mazer CD. Effect of bilateral scalp nerve blocks on postoperative pain and discharge times in patients undergoing supratentorial craniotomy and general anesthesia: a randomized-controlled trial. Can J Anaesth. 2020 Apr;67(4):452-461. doi: 10.1007/s12630-019-01558-7. Epub 2019 Dec 26. PMID 31879855
- [Background] Carella M, Tran G, Bonhomme VL, Franssen C. Influence of Levobupivacaine Regional Scalp Block on Hemodynamic Stability, Intra- and Postoperative Opioid Consumption in Supratentorial Craniotomies: A Randomized Controlled Trial. Anesth Analg. 2021 Feb 1;132(2):500-511. doi: 10.1213/ANE.0000000000005230. PMID 33060491
- [Background] Lamsal R, Rath GP. Pediatric neuroanesthesia. Curr Opin Anaesthesiol. 2018 Oct;31(5):539-543. doi: 10.1097/ACO.0000000000000630. PMID 29985182
- [Background] van Lindert EJ, Liem KD, Geerlings M, Delye H. Bedside placement of ventricular access devices under local anaesthesia in neonates with posthaemorrhagic hydrocephalus: preliminary experience. Childs Nerv Syst. 2019 Dec;35(12):2307-2312. doi: 10.1007/s00381-019-04361-3. Epub 2019 Sep 10. PMID 31506779